CLINICAL TRIAL: NCT00402922
Title: Pericardial Fat and Subclinical and Clinical Measures of Coronary Heart Disease - Ancillary to MESA
Brief Title: Evaluating the Association Between Pericardial Fat and Coronary Heart Disease - Ancillary to MESA
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jingzhong Ding, PhD, Associate Professor, Wake Forest University Health Sciences
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: 1358; R01HL085323-01 (NIH)
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Disease
Keywords: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Coronary heart disease (CHD) is the leading cause of death in the United States. One common risk factor for CHD is obesity. The presence of certain types of fat over others is more commonly associated with the development of CHD. This study will use data from a previous study to examine the association between pericardial fat, a type of fat that surrounds the heart, and CHD.

DETAILED DESCRIPTION:
CHD is caused by a narrowing of the small blood vessels that supply blood and oxygen to the heart. It usually results from atherosclerosis, a condition in which deposits of fat, cholesterol, and other substances build up along the inner walls of arteries. Risk factors for CHD include tobacco use, high blood pressure, diabetes, and obesity. Visceral fat, the type of fat found in the abdomen and surrounding vital organs, is considered a greater risk factor for CHD than subcutaneous fat, the type of fat found directly below the skin. Pericardial fat, the fat surrounding the heart, is similar to visceral fat, and may be particularly damaging because of its lipotoxicity effects and its ability to trigger inflammation in the coronary arteries. Increased amounts of pericardial fat may therefore accelerate the development of atherosclerosis and CHD. The purpose of this study is to evaluate the relationship between pericardial fat and the development of CHD.

This study will use previously collected data from participants in the Multi-Ethnic Study of Atherosclerosis (MESA) study, a study that examined characteristics of the subclinical, or the early stages of, cardiovascular disease in individuals. There will be no study visits specifically for this study. Participants' study data and computed tomography (CT) scans will be analyzed to determine the following: 1) the presence of pericardial fat and subclinical CHD at study entry; 2) changes in pericardial fat levels and plaque formation; and 3) the presence of pericardial fat and CHD at a 6-year follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the MESA study
* Had a baseline and 6-year follow-up CT scan as part of the MESA study

Exclusion Criteria:

* Participant did not have a baseline or 6 year follow-up CT in the MESA study

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participant in the MESA study
Sampling Method: Non-Probability Sample
Enrollment: 6814 (Actual)
Dates: Start 2006-08; Primary Completion 2008-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Coronary heart disease events | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Jingzhong Ding, MD, PhD, Principal Investigator — Wake Forest University Health Sciences